CLINICAL TRIAL: NCT01676766
Title: Novel Quantification Methods for Fundus Flavoprotein Fluorescence and Lipofuscin Fluorescence to Detect Progression in Stargardt Disease
Brief Title: Novel Quantification Methods for Fluorescence to Detect Progression in Stargardt Disease
Status: Terminated | Type: Observational
Why Stopped: Flavoprotein fluorescence machine for the trial is not working so the trial was terminated. No study data was collected prior to termination.
Sponsor: University of Michigan (Other)
Collaborators: Midwest Eye Banks (Other)
Responsible Party: Principal Investigator, K. Thiran Jayasundera, Assistant Professor, Retina and Uveitis, University of Michigan
Other Study IDs: HUM 64388
Record Dates: First submitted 2012-08-23; First posted 2012-08-31 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Stargardt Disease
Keywords: Stargardt Disease; Macular degeneration; Retinal dystrophy
MeSH Terms: conditions — Stargardt Disease; Macular Degeneration; Retinal Dystrophies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to utilize flavoprotein fluorescence and fundus autofluorescence to detect progression of Stargardt macular dystrophy in a pediatric population over the course of a year with the hope of aiding future therapeutic risk-benefit decisions and assessment of outcomes.

Stargardt macular dystrophy is the most common of the juvenile-onset macular dystrophies. Despite determination of ABCA4 as the causative gene, clinicians have been challenged by variability in clinical phenotypes. Given the recent initiation of clinical trials to assess novel treatments (e.g. gene therapy), there is a need to identify patients with the worst prognosis.

The investigators have observed that pediatric patients lose central visual function faster than their adult counterparts. Thus, they present an ideal cohort with which to determine the utility of novel modalities to detect early change. These include flavoprotein fluorescence, a new imaging technique for detecting mitochondrial dysfunction developed at the University of Michigan. Fundus autofluorescence (FAF) is another commonly utilized technique of evaluating hereditary eye diseases. The investigators have developed a novel means of quantifying FAF signatures that will allow documentation of severity as well as detection of progression.

DETAILED DESCRIPTION:
This study will evaluate whether more sophisticated testing and analytic methodologies, including fundus autofluorescence (FAF) and a novel non-invasive method to measure retinal flavoprotein fluorescence (FPF) may be used to better predict Stargardt macular dystrophy progression and monitor treatment effects than conventional modalities such visual acuity and visual field. This method involves the use of novel statistical methods to assess the heterogeneity of fundus autofluorescence images.

Participants will complete 3 visits to the University of Michigan Kellogg Eye Center. Each visit will take approximately 2.5 hours. The initial visit will include a routine clinical eye examination, measurement of best-corrected visual acuity, indirect ophthalmoscopy, microperimetry, frequency-domain optical coherence tomography, Goldmann visual fields, fundus flavoprotein fluorescence (FPF) imaging, and fundus autofluorescence (FAF) and fundus photography. Patients will return for evaluation at 6 and 12 months after their initial visit to repeat testing and imaging.

ELIGIBILITY:
Inclusion Criteria:

* Between the age of 5 and 18 years old
* Clinical diagnosis of Stargardt Disease
* Molecular confirmation of Stargardt Disease (with 2 identified mutations in ABCA4)
* Visual acuity better than 20/100

Exclusion Criteria:

* Limited central vision, defined as visual acuity worse than 20/100
* A diagnosis of any other retinal degenerative disease

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: We will perform an observational clinical study of 25 pediatric patients with Stargardt Disease recruited from the retinal degeneration clinic at the University of Michigan who have two mutations in ABCA4.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2012-09; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pixel intensity quantification of fundus autofluorescence at 6 months | 0 months, 6 months
Change from baseline in pixel intensity quantification of flavoprotein autofluorescence at 6 months | 0 months, 6 months

SECONDARY OUTCOMES:
Change from baseline in pixel intensity quantification of fundus autofluorescence at 12 months | 0 months, 12 months
Change from baseline in pixel intensity quantification of flavoprotein autofluorescence at 12 months | 0 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: K. Thiran Jayasundera, MD, Principal Investigator — University of Michigan Kellogg Eye Center
Locations (1):
- Kellogg Eye Center, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Elner SG, Elner VM, Field MG, Park S, Heckenlively JR, Petty HR. Retinal flavoprotein autofluorescence as a measure of retinal health. Trans Am Ophthalmol Soc. 2008;106:215-22; discussion 222-4. PMID 19277237
- [Background] Field MG, Elner VM, Park S, Hackel R, Heckenlively JR, Elner SG, Petty HR. Detection of retinal metabolic stress resulting from central serous retinopathy. Retina. 2009 Sep;29(8):1162-6. doi: 10.1097/IAE.0b013e3181a3b923. PMID 19491721
- [Background] Field MG, Elner VM, Puro DG, Feuerman JM, Musch DC, Pop-Busui R, Hackel R, Heckenlively JR, Petty HR. Rapid, noninvasive detection of diabetes-induced retinal metabolic stress. Arch Ophthalmol. 2008 Jul;126(7):934-8. doi: 10.1001/archopht.126.7.934. PMID 18625939
- [Background] Chen B, Tosha C, Gorin MB, Nusinowitz S. Analysis of autofluorescent retinal images and measurement of atrophic lesion growth in Stargardt disease. Exp Eye Res. 2010 Aug;91(2):143-52. doi: 10.1016/j.exer.2010.03.021. Epub 2010 Apr 14. PMID 20398653